CLINICAL TRIAL: NCT00190346
Title: Randomized RCT Comparing HH and HME During NIV in Acute Respiratory Failure
Brief Title: Comparison of Humidification Devices During Non Invasive Ventilation, in Acute Respiratory Failure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PHRC 2001
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2005-08

CONDITIONS: Respiratory Failure; COPD; Hypoxemia; Non Invasive Ventilation
Keywords: Acute respiratory distress; with hypercapnia; with hypoxemia; requiring NIV
MeSH Terms: conditions — Respiratory Insufficiency; Pulmonary Disease, Chronic Obstructive; Hypoxia; Acute Lung Injury

INTERVENTIONS:
Device: Humidification devices: HH vs HME

SUMMARY:
Comparison of humidification devices during non invasive ventilation, in acute respiratory failure.

The hypothesis was, due to dead space, lower humidification, a reduced efficiency of the technique (NIV) when HME are used in comparison with HH.

DETAILED DESCRIPTION:
Comparison of humidification devices during non invasive ventilation, in acute respiratory failure.

The hypothesis was, due to dead space, lower humidification, a reduced efficiency of the technique (NIV) when HME are used in comlparison with HH Several physiological previously performed showed that 1) with HME, because of its working principles, humidification was reduced because of leaks 2) work of breathing was increased with HME because of dead space and 3) alveolar ventilation was reduced with HME because of additional technical dead space.

For these reasons, the hypothesis was an improvement of NIV tolerance, of efficiency to clear te CO2 with HH in comparison with HME and finally to reduce the intubation rate with HH.

The patients were included when requiring NIV (see inclusion and exclusion criteria) and randomisation was performed with stratification according to presence or absence of respiratory acidosis.

The number of patients to include was baszd on the hypothesis that intubation rate would be reduced from 40 with HME to 25% with HME. A total of 250 patients was required with alpha risk of 0,05 and beta risk of 0,2 (power 80%). Intubation criteria were predefined according to the litterature. The expected duration was 18 months. The official support was institutional (DRRC of AP-HP). HH were furnished free of charge, as well as HME. Masks used were the same in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years
* Exacerbation of dyspnea lasting less than two weeks

TWO OR THREE following criteria :

* Respiratory rate higher or equal to 25 b/min
* SaO2 lower or equal to 90% (breathing room air or oxygen)
* Arterial pH < 7.35

Exclusion Criteria:

* immediate need for intubation
* cardiac arrest or RR< 10 breaths/min.
* systemic hypotension (SAP < 80 mmHg ) with no response to 500 ml of macromolecules
* coma defined by GCS < 8.
* high probability of surgical procedure
* major facial deformity
* pneumothorax
* bad short-term prognosis
* refusal of intubation by the patient or do not intubated order.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2001-12; Study Completion 2003-04

PRIMARY OUTCOMES:
Intubation rate | during the study

SECONDARY OUTCOMES:
-Physiological outcome at 1,3 and 6 hours (arterial blood gases, respiratory rate) | during the study
-Intolerance of NIV | during the study
- Frequency of VAP | during the study
- Duration of total MV duration | during the study
- ICU LOS | during the study
- Hospital LOS | during the study
- Mortality (ICU and hospital) | during the study

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Best, Study Chair — DRRC hopitaux de Paris
Locations (14):
- Département d'Anesthésie - Hôpital de l'Enfant Jésus, Québec, Quebec, Canada
- France (11):
  - Hôpital Victor Dupouy, Argenteuil, Argenteuil
  - CHU de La Cavale Blanche, Brest
  - Réanimation du Service de Pneumologie - Centre Hospitalier Beaujon, Clichy
  - Réanimation Médicale - Hôpital Louis Mourier, Colombes
  - Département d'Anesthésie-Réanimation "B" - CHU Saint Eloi, Montpellier
  - Hôpital Georges Pompidou HEGP, Paris
  - Réanimation du Service Pneumologie - Hôtel Dieu, Paris
  - Réanimation pneumologique, Hôpital Pitié Salpétrière, Paris
  - Réanimation Pneumologique- CHU Tenon, Paris
  - Réanimation Médicale - Centre Hospitalier Intercommunal de Poissy, Poissy
  - Réanimation Médicale, Hôpital Charles Nicolle, Rouen
- Istituto di anestesiologia e Rianimazione - Università Cattolica Policlinico A. Gemelli, Roma, Italy
- Réanimation Polyvalente - CHU Fatima Bourguiba, Monastir, Tunisia

REFERENCES:
- [Derived] Lellouche F, L'Her E, Abroug F, Deye N, Rodriguez PO, Rabbat A, Jaber S, Fartoukh M, Conti G, Cracco C, Richard JC, Ricard JD, Mal H, Mentec H, Loisel F, Lacherade JC, Taille S, Brochard L. Impact of the humidification device on intubation rate during noninvasive ventilation with ICU ventilators: results of a multicenter randomized controlled trial. Intensive Care Med. 2014 Feb;40(2):211-219. doi: 10.1007/s00134-013-3145-z. Epub 2013 Nov 26. PMID 24275900